CLINICAL TRIAL: NCT05611268
Title: Pentoxifylline as an Adjunct Therapy for Patients With Eisenmenger Syndrome: a Randomized Study
Brief Title: Pentoxifylline as an Adjunct Therapy for Patients With Eisenmenger Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: InCor Heart Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: CAAE 57562322.5.0000.0068
Record Dates: First submitted 2022-08-24; First posted 2022-11-10 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Eisenmenger Syndrome
Keywords: Pulmonary Hypertension; Congenital Heart Disease; Thrombosis; Pentoxifylline; Thrombomodulin; Tissue Factor
MeSH Terms: conditions — Eisenmenger Complex; Hypertension, Pulmonary; Heart Defects, Congenital; Thrombosis | interventions — Pentoxifylline

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The professional responsible for obtainment of laboratory data including outcome measures will not have access to any clinical data or patient allocation to the study groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- No treatment group (No Intervention): 24 patients that will continue receiving routine treatment for PAH
- Pentoxifylline (Other): 24 patients that will receive pentoxifylline and the routine treatment for PAH
  Interventions: Drug: Pentoxifylline

INTERVENTIONS:
Drug: Pentoxifylline — Oral Pentoxifylline 400 mg/day for 30 days, followed by 800 mg/day for 150 days
  Arms: Pentoxifylline

SUMMARY:
The Eisenmenger syndrome corresponds to the most advanced form of pulmonary arterial hypertension associated with congenital heart disease. The syndrome causes chronic hypoxemia, with an increase in erythrocyte mass, which predisposes to thrombotic complications. Pentoxifylline is a xanthine derivative and it is considered as a hemorrheological agent with described effects of reduction in erythrocyte and platelet aggregation, adhesion and activation of leukocytes, and endothelial damage. The main objective of this study is to verify if the chronic oral administration of pentoxifylline to Eisenmenger patients induces an increase in the circulating levels of thrombomodulin, a naturally occurring proteoglycan with anticoagulant, anti thrombotic and anti-inflammatory properties.

DETAILED DESCRIPTION:
The Eisenmenger syndrome corresponds to the most advanced form of pulmonary arterial hypertension associated with congenital heart disease. The syndrome causes chronic hypoxemia, with an increase in erythrocyte mass, which predisposes to thrombotic complications. It also involves endothelial dysfunction characterized by increase in the circulating levels of von Willebrand factor, tissue-type plasminogen activator and P-selectin, with a reduction in the plasma concentration of thrombomodulin. The usual drug treatment is represented by the use of prostanoids, endothelin receptor antagonists, phosphodiesterase-5 inhibitors and, eventually, anticoagulation with warfarin. However, the difficulty of controlling the chronic use of warfarin and the few studies with other oral anticoagulants, brings the possibility of using drugs not specifically designated as coagulation inhibitors, such as pentoxifylline. This drug is a xanthine derivative and it is considered as a hemorrheological agent with described effects of reduction in erythrocyte and platelet aggregation, adhesion and activation of leukocytes, and endothelial damage. It is, therefore, considered as an agent capable of reducing blood viscosity and improving erythrocyte deformability probably due to an increase in intracellular adenosine triphosphate (ATP), with a reduction in Ca++ and phosphorylation of membrane proteins. The objective of this study is to verify if the chronic oral administration of pentoxifylline: 1) induces an increase in the circulating levels of thrombomodulin, a naturally occurring proteoglycan with anticoagulant, anti thrombotic and anti-inflammatory properties; 2) stabilizes or induces a reduction in circulating tissue factor and thrombin-antithrombin complexes; 3) changes the expression of thrombomodulin and tissue factor in circulating monocytes; 4) offers protection against the occurrence of predefined clinical events; 5) provides improvement in physical capacity, peripheral oxygen saturation, hematocrit level and right ventricular function. The main study outcome is biochemical: change from baseline (increase) in circulating levels of thrombomodulin at 3 months and 6 months of oral use of pentoxifylline. It will be a prospective, single-center, randomized study. Forty-eight adult patients with Eisenmenger syndrome who are already using specific therapies for pulmonary arterial hypertension will be included and these will be randomized to receive pentoxifylline as an adjunctive treatment or remain under routine therapeutic measures for pulmonary arterial hypertension. Oral pentoxifylline will be started at the dose of 400 mg/day for 30 days, followed by 800 mg/day for 5 months, completing the 6-month period of the study. The routine treatment for pulmonary arterial hypertension will be maintained for all patients.

ELIGIBILITY:
Inclusion Criteria:

1. Eisenmenger syndrome in functional class II, III or IV (World Health Organization for Pulmonary Hypertension).
2. Using or not oral anticoagulation with warfarin.

Exclusion Criteria:

1. Hospitalized.
2. History of relevant and/or repetitive bleeding.
3. Relevant comorbidities with specific treatments.
4. Systemic syndromes, except Down syndrome.
5. Candidates for surgical treatment of any nature, except dental.
6. Clinically manifest systemic infectious or inflammatory disease.
7. Thrombocytopenia (<80x10*9 platelets/L).
8. Patients in chronic anticoagulation regimen other than warfarin.
9. Diabetics individuals.
10. Pregnancy in progress, interruption of contraception or amenorrhea.
11. History of intolerance of pentoxifylline or other xanthine derivatives.
12. "Creatinine clearance" less than or equal to 30 mL/minute.

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-06-03 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Plasma concentration of Thrombomodulin | 3 months and 6 months
  Change in plasma concentration of thrombomoduin at 3 months and 6 months of pentoxifylline therapy compared to baseline.

SECONDARY OUTCOMES:
Plasma concentration of tissue factor | 3 months and 6 months
  Change in plasma concentration of tissue factor at 3 months and 6 months of pentoxifylline therapy compared to baseline.
Monocyte thrombomodulin content | 3 months and 6 months
  Change in mean fluorescence intensity (MFI) for thrombomodulin in circulating (blood) monocytes measured by flow cytometry 3 months and 6 months of pentoxifylline therapy compared to baseline.
Monocyte tissue factor content | 3 months and 6 months
  Change in mean fluorescence intensity (MFI) for tissue factor in circulating (blood) monocytes measured by flow cytometry 3 months and 6 months of pentoxifylline therapy compared to baseline.
Plasma concentration of other markers of thrombosis | 3 months and 6 months
  Change in plasma concentration of D-dimer and thrombin-antithrombin complexes at 3 months and 6 months of pentoxifylline therapy compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Augusto Barbosa Lopes, MD, Principal Investigator — InCor Heart Institute
Locations (1):
- Antonio Augusto Barbosa Lopes, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No